CLINICAL TRIAL: NCT03911778
Title: Prospective Study of the Evolution of Symptoms After Sacrospinofixation With Posterior Isthmic Band
Brief Title: Evolution of Symptoms After Sacrospinofixation With Posterior Isthmic Band
Acronym: SPIP
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0256; 2019-A01044-53 (Other: ID-RCB)
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-01

CONDITIONS: Apical Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sacrospinofixation: Patients with apical symptomatic prolapse ≥ II in the POP-Q classification and for whom sacrospinofixation with posterior isthmic BSC Mesh is planned
  Interventions: Other: Improvement of symptoms

INTERVENTIONS:
Other: Improvement of symptoms — Improvement of symptoms on the Patient Global Impression of Improvement Index (PGI-I) scale (score 1, 2, or 3) at 6 weeks postoperatively

SUMMARY:
Prolapse is a condition that can cause disabling pelvic, urinary or sexual function disorders and impaired quality of life.

Regarding the prolapse of the middle floor, the vaginal sacrospinofixation according to Richter is the reference technique for the suspension of the vaginal fundus. But the technique of sacrospinofixation vaginally is not without several difficulties in the short term but also in the medium and long term.

Recently, anchoring devices have been developed to limit the dissection of the sacrospinous ligament and the operative exposure by the sometimes traumatic valves.

The investigating team uses a technical variant in the form of an isthmic posterior strip of light weight and whose arms are sutured to the sacrospinous ligaments. The advantages of this isthmic strip are based on its small size, its very low basis weight and its wide mesh (improvement of tolerance) via a mini-invasive vaginal approach (thus allowing ambulatory care).

Patient functional discomfort is the main problem related to the presence of a prolapse, therefore, the researchers wish to evaluate patient feelings following the use of this isthmic band. The researchers' hypothesis is that the sacrospinofixation technique with posterior isthmic band Bilateral Sacrospinous Colposuspension (BSC) Mesh (Agency for Medical Innovations (AMI) laboratory) improves symptoms experienced by patients with mid-level prolapse.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* apical prolapse requiring surgical correction of grade II or greater in the Pelvic Organ Prolapse Quantification (POP-Q) classification
* patients who wish an intervention because of the discomfort caused by prolapse
* sacrospinofixation procedure with posterior isthmic band Bilateral Sacrospinous Colposuspension (BSC) Mesh provided
* person having expressed his non-opposition

Exclusion Criteria:

* apical prolapse of stage < II in the Pelvic Organ Prolapse Quantification (POP-Q) classification, and prolapse without functional discomfort
* disorders leading to an unacceptable risk of postoperative complications sought during the interrogation of the patient (disorders of blood coagulation, disorders of the immune system, progressive diseases ....)
* reduced mobility of the lower limbs (not allowing positioning for surgery)
* pregnancy or any plans for pregnancy during the study period
* evolutionary or latent infection
* known hypersensitivity to polypropylene
* inability to understand the information given
* person deprived of liberty, under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with apical symptomatic prolapse ≥ II in the Pelvic Organ Prolapse Quantification (POP-Q) classification and for whom sacrospinofixation with posterior isthmic Bilateral Sacrospinous Colposuspension (BSC) Mesh is planned
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Improvement of symptoms | 6 weeks postoperatively
  Percentage of patients with improvement of their symptoms on the Patient Global Impression of Improvement Index (PGI-I) scale (score 1, 2, or 3)

CONTACTS AND LOCATIONS:
Overall Officials: Gautier CHENE, Ph.D., Principal Investigator — Hospices Civils de Lyon, Hôpital Femme Mère Enfant
Locations (1):
- Service de gynecologie Hôpital Femme mère enfant, Bron, France